CLINICAL TRIAL: NCT05047874
Title: Comparison of High-dose, Short-term Steroid and Low-dose Long-term Steroid Use in ARDS Caused by COVID-19 - Retrospective Cross-sectional Study
Brief Title: High-dose, Short-term Steroid and Low-dose Long-term Steroid Use in ARDS Caused by COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, IKUPELI, investigator, Biruni University
Other Study IDs: BIRUNI 1
Record Dates: First submitted 2021-09-16; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Short-term (3 Days) High-dose (1000 mg) Systemic Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- short-term (3 days) high-dose (1000 mg) systemic methylprednisolone: retrospectively, the 15-day continuous hemodynamic, laboratory and clinical course of COVID 19 patients to whom we administered short-term (3 days) high-dose (1000 mg) systemic methylprednisolone
  Interventions: Behavioral: systemic methylprednisolone
- low-dose long-term (2x 40 mg) systemic methylprednisolone: retrospectively, the 15-day continuous hemodynamic, laboratory and clinical course of COVID 19 patients to whom low-dose long-term (2x 40 mg) systemic methylprednisolone
  Interventions: Behavioral: systemic methylprednisolone

INTERVENTIONS:
Behavioral: systemic methylprednisolone — short-term (3 days) high-dose (1000 mg) systemic methylprednisolone and low-dose long-term (2x 40 mg) systemic methylprednisolone

SUMMARY:
In this study, we aimed to compare, retrospectively, the 15-day continuous hemodynamic, laboratory and clinical course of COVID 19 patients to whom we administered short-term (3 days) high-dose (1000 mg) systemic methylprednisolone with those to whom low-dose long-term (2x 40 mg) systemic methylprednisolone was administered.

ELIGIBILITY:
Inclusion Criteria:

* Between June 1, 2020 and February 1, 2021, hospitalized in the General intensive care unit of Biruni University Medical Faculty Hospital with the diagnosis of COVID 19;
* patients over 18 years of age; (for the diagnosis of COVID 19; Identification of SARS-CoV-2 by reverse transcription-polymerase chain reaction (RT-PCR) in nasopharyngeal swab or sputum samples and Abnormal lung computed tomography finding (CT) scan finding with <90% oxygen saturation at rest (bilateral, subpleural, peripheral ground glass opacities)

Exclusion Criteria:

* Patients with a diagnosis of steroid allergy or developing during treatment;
* pregnant or lactating women;
* Patients with active malignancy;
* Patients taking any immunosuppressive agent.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: File records of patients over the age of 18 who were admitted to the General intensive care unit of Biruni University Medical Faculty Hospital between 1 June 2020 and 1 February 2021 with the diagnosis of COVID 19
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
C Reaktif Protein | 15 DAYS
  level of C Reaktif Protein

CONTACTS AND LOCATIONS:
Locations (1):
- Ilke Kupeli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Buttgereit F, Straub RH, Wehling M, Burmester GR. Glucocorticoids in the treatment of rheumatic diseases: an update on the mechanisms of action. Arthritis Rheum. 2004 Nov;50(11):3408-17. doi: 10.1002/art.20583. No abstract available. PMID 15529366
- [Result] Rodriguez-Molinero A, Perez-Lopez C, Galvez-Barron C, Minarro A, Rodriguez Gullello EA, Collado Perez I, Mila Rafols N, Monaco EE, Hidalgo Garcia A, Ananos Carrasco G, Chamero Pastilla A; group of researchers for COVID-19 of the Consorci Sanitari de l'Alt Penedes i Garraf (CSAPG). Association between high-dose steroid therapy, respiratory function, and time to discharge in patients with COVID-19: Cohort study. Med Clin (Engl Ed). 2021 Jan 10;156(1):7-12. doi: 10.1016/j.medcle.2020.08.001. Epub 2020 Nov 27. PMID 33263084
- [Result] Edalatifard M, Akhtari M, Salehi M, Naderi Z, Jamshidi A, Mostafaei S, Najafizadeh SR, Farhadi E, Jalili N, Esfahani M, Rahimi B, Kazemzadeh H, Mahmoodi Aliabadi M, Ghazanfari T, Sattarian M, Ebrahimi Louyeh H, Raeeskarami SR, Jamalimoghadamsiahkali S, Khajavirad N, Mahmoudi M, Rostamian A. Intravenous methylprednisolone pulse as a treatment for hospitalised severe COVID-19 patients: results from a randomised controlled clinical trial. Eur Respir J. 2020 Dec 24;56(6):2002808. doi: 10.1183/13993003.02808-2020. Print 2020 Dec. PMID 32943404
- [Result] Li J, Liao X, Zhou Y, Wang L, Yang H, Zhang W, Zhang Z, Kang Y. Comparison of Associations Between Glucocorticoids Treatment and Mortality in COVID-19 Patients and SARS Patients: A Systematic Review and Meta-Analysis. Shock. 2021 Aug 1;56(2):215-228. doi: 10.1097/SHK.0000000000001738. PMID 33555845